CLINICAL TRIAL: NCT00976911
Title: AURELIA: A Multi-center, Open-label, Randomised, Two-arm Phase III Trial of the Effect on Progression Free Survival of Bevacizumab Plus Chemotherapy Versus Chemotherapy Alone in Patients With Platinum-resistant, Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: AURELIA: A Study of Avastin (Bevacizumab) Added to Chemotherapy in Patients With Platinum-resistant Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO22224; 2009-011400-33 (EudraCT Number)
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2015-02-25 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; liposomal doxorubicin; Paclitaxel; Topotecan

ARMS (2):
- Chemotherapy (Active Comparator): Participants received one of the following chemotherapies at the discretion of the investigator: paclitaxel, 80 milligrams per square meter (mg/m^2) as a 1-hour intravenous (IV) infusion on Days 1, 8, 15, and 22 every 4 weeks (q4w) OR topotecan 4 mg/m^2 as a 30-minute IV infusion on Days 1, 8, and 15 q4w (alternatively, a 1.25 mg/m^2 dose could have been administered over 30 minutes on Days 1-5 every 3 weeks [q3w]) OR pegylated liposomal doxorubicin (PLD) 40 mg/m^2 as a 1 milligram per minute (mg/min) infusion on Day 1 q4w (after Cycle 1 the drug could have been administered as a 1 hour infusion). Depending on chosen chemotherapy, pre-medication was implemented according to local practices.
  Interventions: Drug: liposomal doxorubicin; Drug: paclitaxel; Drug: topotecan
- Chemotherapy + Bevacizumab (Experimental): Participants received one of the following chemotherapies at the discretion of the investigator: paclitaxel, 80 mg/m^2 as a 1-hour IV infusion on Days 1, 8, 15, and 22 q4w OR topotecan 4 mg/m^2 as a 30-minute IV infusion on Days 1, 8, and 15 q4w (alternatively, a 1.25 mg/m^2 dose could have been administered over 30 minutes on Days 1-5 q3w) OR PLD 40 mg/m^2 as a 1 mg/min infusion on Day 1 q4w (after Cycle 1 the drug could have been administered as a 1 hour infusion. Depending on chosen chemotherapy, pre-medication was implemented according to local practices. The chosen chemotherapy was combined with bevacizumab 10 milligrams per kilogram (mg/kg) IV every 2 weeks (q2w; or bevacizumab 15 mg/kg q3w if used in combination with topotecan 1.25 mg/m^2 on Days 1-5 on a q3w schedule). The initial bevacizumab infusion was over 90 minutes, with subsequent infusions over 60 minutes and then 30 minutes, as tolerated.
  Interventions: Drug: Bevacizumab; Drug: liposomal doxorubicin; Drug: paclitaxel; Drug: topotecan

INTERVENTIONS:
Drug: Bevacizumab — 10m/kg iv every 2 weeks or 15mg/kg iv every 3 weeks
  Other Names: Avastin
  Arms: Chemotherapy + Bevacizumab
Drug: liposomal doxorubicin — 40mg/m2 iv every 4 weeks
Drug: paclitaxel — 80mg/m2 iv on days 1, 8, 15 and 22 of each 4-week cycle
Drug: topotecan — 4mg/m2 iv on days 1, 8 and 15 of each 4-week cycle, or 1.25 mg/kg on days 1-5 of each 3-week cycle

SUMMARY:
This randomized, open-label, 2-arm study will evaluate the efficacy and safety of Avastin added to chemotherapy versus chemotherapy alone in patients with epithelial ovarian, fallopian tube or primary peritoneal cancer with disease progression within 6 months of platinum therapy. All patients will receive standard chemotherapy with either paclitaxel or topotecan or liposomal doxorubicin. Patients randomized to Arm 2 of the study will receive Avastin (10 mg/kg iv 2-weekly or 15 mg/kg iv 3-weekly) concomitantly. Anticipated time on study treatment is until disease progression. Patients will then receive standard of care, those in Arm 1 (chemotherapy only) may opt to receive Avastin (15 mg/kg iv 3-weekly). Target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >/=18 years of age
* epithelial ovarian, fallopian tube or primary peritoneal cancer
* platinum-resistant disease (disease progression within <6 months of platinum therapy)
* EOCG performance status of 0-2

Exclusion Criteria:

* non-epithelial tumours
* ovarian tumours with low malignant potential
* previous treatment with >2 chemotherapy regimens
* prior radiotherapy to the pelvis or abdomen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2009-10-29 (Actual); Primary Completion 2014-07-09 (Actual); Study Completion 2014-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (117):
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
  - Clinique Ste-Elisabeth, Namur
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo
  - University Clinical Center Tuzla; Clinic for Gynecology and Obstetrition, Tuzla
- Denmark (4):
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Regionshospitalet Herning; Onkologisk afdeling, Herning
  - Rigshospitalet; Onkologisk Klinik, København Ø
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital; Gynaecology & Obstetrics Dept, Oulu
- France (36):
  - Clinique Sainte Catherine; Hopital De Semaine, Avignon
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Institut Bergonie; Gynecologie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Ch De Brive La Gaillarde; Radiotherapie Oncologie, Brive-la-Gaillarde
  - Centre Francois Baclesse; Urologie Gynecologie, Caen
  - Centre Jean Perrin; Hopital De Jour, Clermont-Ferrand
  - Hopital Louis Pasteur; Medecine B, Colmar
  - Institut Daniel Hollard; Chimiotherapie Ambulatoire, Grenoble
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Hopital La Source; Onco Med Hematologie Clinique, La Source
  - Hopital Andre Mignot; Hematologie - Oncologie, Le Chesnay
  - Centre Jean Bernard, Le Mans
  - Centre Oscar Lambret; Cancerologie Gynecologique, Lille
  - Clin Mut De Lyon Eugene Andre; Medecine 3 A, Lyon
  - Hopital Layne; Medecine Ambulatoire, Mont-de-Marsan
  - Centre Val Aurelle Paul Lamarque; Medecine A1 A2, Montpellier
  - Polyclinique Gentilly; CHIMIOTHERAPIE AMBULATOIRE, Nancy
  - Centre Catherine de Sienne; Chimiotherapie, Nantes
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Polyclinique Kenval ; Radiotherapie Oncologie, Nîmes
  - Hotel Dieu; Hematologie- Oncologie, Paris
  - Institut Curie; Oncologie Medicale, Paris
  - Hopital Saint Louis ; Service d Oncologie Medicale Fougere 6 (Pr Misset), Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Clinique Francheville; Radiotherapie, Périgueux
  - Institut Jean Godinot; Oncologie Medicale, Reims
  - Centre Henri Becquerel; Oncologie Medicale, Rouen
  - Clinique Armoricaine Radiologie; Cons Externes, Saint-Brieuc
  - Centre Rene Huguenin; Medecine B, Saint-Cloud
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Centre Radiotherapie Etienne Dolet, Saint-Nazaire
  - Hopital Civil; Expl Fonct Systeme Nerveux, Strasbourg
  - Hopitaux Du Leman Site Thonon; Maternite Gynecologie, Thonon-les-Bains
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
- Germany (26):
  - HELIOS Klinikum Berlin-Buch; Klinik für Gynäkologie und Geburtshilfe, Berlin
  - Campus Virchow-Klinikum Charité; Centrum 17; Klinik für Gynäkologie, Berlin
  - Evangelischen Krankenhauses Düsseldorf; Frauenklinik, Düsseldorf
  - Uni-Frauenklinik, Düsseldorf
  - Universitätsklinikum Erlangen; Frauenklinik, Erlangen
  - Universitätsklinikum Essen; Zentrum Für Frauenheilkunde, Essen
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Klinik für Frauenheilkunde und Geburtshilfe, Frankfurt
  - Kath.Marienkrankenhaus gGmbH Frauenklinik, Hamburg
  - Gynaekologisch-Onkologische Schwerpunktpraxis Prof. Dr. med. Lueck, Dr. Schrader und Dr. Noeding, Hanover
  - Praxisgemeinschaft; Frauenärzte am Bahnhofsplatz, Hildesheim
  - Klinikum Kassel GmbH; Klinik für Frauenheilkunde und Geburtshilfe, Kassel
  - UNI-Klinikum Campus Kiel Klinik für Gynäkologie und Geburtshilfe, Kiel
  - HELIOS Klinikum Krefeld; Klinik für Frauenheilkunde und Geburtshilfe, Krefeld
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Universitätsklinikum Mannheim; Frauenklinik, Mannheim
  - Klinikum der Universität München; Campus Großhadern; Klinik und Poliklinik für Frauenheilkunde, München
  - Klinikum Nord Frauenklinik, Nuremberg
  - Sana Klinikum Offenbach GmbH; Klinik für Gynäkologie & Geburtshilfe, Offenbach
  - Oncologianova GmbH, Recklinghausen
  - Universitätsfrauen- und Poliklinik am Klinikum Suedstadt, Rostock
  - Städtisches Klinikum Solingen; Klinik für Frauenheilkunde und Geburtshilfe, Solingen
  - Robert-Bosch-Krankenhaus; Interdisziplinäres Zentrum; Tumorzentrum, Stuttgart
  - Universitätsklinik Tübingen; Frauenklinik & Poliklinik, Tübingen
  - Universitätsklinikum Ulm Am Michelsberg; Frauenklinik, Ulm
  - Dr. Horst-Schmidt-Kliniken; Frauenheilkunde & Geburtshilfe, Wiesbaden
- University Hospital of Alexandra, Athens, Greece
- Italy (8):
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia, Udine, Friuli Venezia Giulia
  - AZIENDA POLICLINICO UMBERTO I; Ginecologia ed Ostetricia, Rome, Lazio
  - Istituto Regina Elena; Oncologia Medica A, Rome, Lazio
  - Ospedale S.G.Calibita Fatebenefratelli; Unità Operativa Oncologia, Rome, Lazio
  - Ospedali Riuniti; Divisione Ostetricia e Ginecologia, Bergamo, Lombardy
  - Az. Osp. Carlo Poma; Divisione Di Oncologia Medica, Mantova, Lombardy
  - Istituto Nazionale dei Tumori; Divisione Oncologia Chirurgica e Ginecologica, Milan, Lombardy
- Netherlands (6):
  - Meander Mc, Locatie Lichtenberg; Dept of Lung Diseases, Amersfoort
  - Catharina ZKHS; Inwendige Geneeskunde Afd., Eindhoven
  - Martini Ziekenhuis; Dept of Internal Medicine, Groningen
  - Stichting St. Antonius Ziekenhuis, Nieuwegein
  - Leyenburg Ziekenhuis; Internal Medecine, The Hague
  - Universitair Medisch Centrum Utrecht; Inwendige Geneeskunde Afd., Utrecht
- Norway (2):
  - The Norvegian Radium Hospital Montebello; Dept of Oncology, Oslo
  - St. Olavs Hospital; Kvinneklinikken, Trondheim
- Portugal (2):
  - IPO de Lisboa; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Spain (15):
  - Hospital Son Llatzer; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital de Terrassa; Servicio de Oncologia, Barcelona
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Centro Oncologico MD Anderson Internacional; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Oncologia, Murcia
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (4):
  - Uni Hospital Linkoeping; Dept. of Oncology, Linköping
  - Örebro University Hospital; Department of Gynecologic Oncology, Örebro
  - Norrlands Uni Hospital; Onkologi Avd., Umeå
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Turkey (Türkiye) (4):
  - Adana Baskent University Hospital; Medical Oncology, Adana
  - Ankara Baskent University Medicine Faculty; Gynaecology, Ankara
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - Anadolu Health Center; Medical Oncology, Kocaeli

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Roncolato FT, Gibbs E, Lee CK, Asher R, Davies LC, Gebski VJ, Friedlander M, Hilpert F, Wenzel L, Stockler MR, King M, Pujade-Lauraine E. Quality of life predicts overall survival in women with platinum-resistant ovarian cancer: an AURELIA substudy. Ann Oncol. 2017 Aug 1;28(8):1849-1855. doi: 10.1093/annonc/mdx229. PMID 28595285
- [Derived] Bamias A, Gibbs E, Khoon Lee C, Davies L, Dimopoulos M, Zagouri F, Veillard AS, Kosse J, Santaballa A, Mirza MR, Tabaro G, Vergote I, Bloemendal H, Lykka M, Floquet A, Gebski V, Pujade-Lauraine E. Bevacizumab with or after chemotherapy for platinum-resistant recurrent ovarian cancer: exploratory analyses of the AURELIA trial. Ann Oncol. 2017 Aug 1;28(8):1842-1848. doi: 10.1093/annonc/mdx228. PMID 28481967
- [Derived] Sorio R, Roemer-Becuwe C, Hilpert F, Gibbs E, Garcia Y, Kaern J, Huizing M, Witteveen P, Zagouri F, Coeffic D, Luck HJ, Gonzalez-Martin A, Kristensen G, Levache CB, Lee CK, Gebski V, Pujade-Lauraine E; AURELIA Investigators. Safety and efficacy of single-agent bevacizumab-containing therapy in elderly patients with platinum-resistant recurrent ovarian cancer: Subgroup analysis of the randomised phase III AURELIA trial. Gynecol Oncol. 2017 Jan;144(1):65-71. doi: 10.1016/j.ygyno.2016.11.006. Epub 2016 Nov 18. PMID 27871723
- [Derived] Stockler MR, Hilpert F, Friedlander M, King MT, Wenzel L, Lee CK, Joly F, de Gregorio N, Arranz JA, Mirza MR, Sorio R, Freudensprung U, Sneller V, Hales G, Pujade-Lauraine E. Patient-reported outcome results from the open-label phase III AURELIA trial evaluating bevacizumab-containing therapy for platinum-resistant ovarian cancer. J Clin Oncol. 2014 May 1;32(13):1309-16. doi: 10.1200/JCO.2013.51.4240. Epub 2014 Mar 31. PMID 24687829
- [Derived] Pujade-Lauraine E, Hilpert F, Weber B, Reuss A, Poveda A, Kristensen G, Sorio R, Vergote I, Witteveen P, Bamias A, Pereira D, Wimberger P, Oaknin A, Mirza MR, Follana P, Bollag D, Ray-Coquard I. Bevacizumab combined with chemotherapy for platinum-resistant recurrent ovarian cancer: The AURELIA open-label randomized phase III trial. J Clin Oncol. 2014 May 1;32(13):1302-8. doi: 10.1200/JCO.2013.51.4489. Epub 2014 Mar 17. PMID 24637997

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Started | 182 | 179
Completed | 0 (At time of clinical cutoff for overall survival and safety (25 January 2013)) | 0 (At time of clinical cutoff for overall survival and safety (25 January 2013))
Not Completed | 182 | 179
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Death | 138 | 126
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Other | 8 | 9
Not completed — In Follow-Up as of 25 Jan 2013 | 30 | 37

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Chemotherapy: Participants received one of the following chemotherapies at the discretion of the investigator: paclitaxel, 80 mg/m^2 as a 1-hour IV infusion on Days 1, 8, 15, and 22 q4w OR topotecan 4 mg/m^2 as a 30-minute IV infusion on Days 1, 8, and 15 q4w (alternatively, a 1.25 mg/m^2 dose could have been administered over 30 minutes on Days 1-5 q3w) OR PLD 40 mg/m^2 as a 1 mg/min infusion on Day 1 q4w (after Cycle 1 the drug could have been administered as a 1 hour infusion). Depending on chosen chemotherapy, pre-medication was implemented according to local practices.
- Chemotherapy + Bevacizumab: Participants received one of the following chemotherapies at the discretion of the investigator: paclitaxel, 80 mg/m^2 as a 1-hour IV infusion on Days 1, 8, 15, and 22 q4w OR topotecan 4 mg/m^2 as a 30-minute IV infusion on Days 1, 8, and 15 q4w (alternatively, a 1.25 mg/m^2 dose could have been administered over 30 minutes on Days 1-5 q3w) OR PLD 40 mg/m^2 as a 1 mg/min infusion on Day 1 q4w (after Cycle 1 the drug could have been administered as a 1 hour infusion). Depending on chosen chemotherapy, pre-medication was implemented according to local practices. The chosen chemotherapy was combined with bevacizumab 10 mg/kg IV q2w (or bevacizumab 15 mg/kg q3w if used in combination with topotecan 1.25 mg/m^2 on Days 1-5 on a q3w schedule). The initial bevacizumab infusion was over 90 minutes, with subsequent infusions over 60 minutes and then 30 minutes, as tolerated.
- Total: Total of all reporting groups
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab | Total
Number analyzed (Participants) | 182 | 179 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.8) | 60.0 (11.1) | 60.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 179 | 361
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death (Data Cutoff 14 November 2011)
Description: Progression free survival was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurs first. Progression was based on tumour assessment made by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria (for participants with measurable disease), and for those with non-measurable disease presence or absence of lesions was noted.
Time Frame: Screening Visit, Every 8 weeks (or 9 weeks if receiving topotecan) until progression reported between day of first participant randomized (29 October 2009) until cutoff date of 14 November 2011
Population: ITT Population: All participants randomized to study treatment, irrespective of whether or not the assigned treatment was actually received. For all efficacy analyses, participants were grouped according to the treatment assigned at randomization
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 182 | 179
percentage of participants | 92.3 | 78.8

2. Secondary Outcome: Percentage of Participants With Best Overall Confirmed Objective Response of Complete Response (CR) or Partial Response (PR) Per Modified RECIST (Data Cutoff 14 November 2011)
Description: Objective Response was determined by the investigator using modified RECIST criteria, Version 1.0. An objective response was a complete or partial overall confirmed response as determined by investigators. CR defined as complete disappearance of all target and non-target lesions and no new lesions. PR defined as greater than or equal to (≥) 30 percent (%) decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions. 95% CI computed using the normal approximation to the binomial distribution.
Time Frame: as for outcome 1
Population: ITT Population; only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 144 | 142
percentage of participants | 12.5 [7.1 to 17.9] | 28.2 [20.8 to 35.6]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; Difference in Response Rates = 15.7, 95% CI 2-sided [6.5 to 24.8]
Statistical Analysis 2: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.0010, Pearson's chi-square; unstratified analysis
Statistical Analysis 3: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel — Stratified analysis: The strata were chemotherapy selected (paclitaxel, PLD, or topotecan), prior anti-angiogenic therapy (yes or no), and platinum-free interval (<3 or 3-6 months)

3. Secondary Outcome: Duration of Objective Response (Data Cutoff 14 November 2011)
Description: For randomized participants who achieved an objective response per modified RECIST, duration of objective response was defined as the time from the date of the first occurrence of a CR or PR (whichever occurred first) until the date that progressive disease or death was documented (whichever occurred first). Participants who had an objective response and did not experience disease progression or death by the time of analysis were censored at the time of the last tumor assessment. Summaries of duration of objective response (median and percentiles) were estimated from Kaplan-Meier curves. 95% CI for duration of objective response was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: ITT Population; only participants with a best overall confirmed response of CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 18 | 40
months | 5.4 [3.81 to 9.23] | 9.4 [6.60 to 11.63]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.0202, Log Rank — Unstratified analysis; Hazard Ratio (HR) = 0.450, 95% CI 2-sided [0.225 to 0.900] — Hazard ratio was estimated by unstratified Cox regression model
Statistical Analysis 2: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.0081, Peto-Peto-Prentice

4. Secondary Outcome: Percentage of Participants Who Died (Data Cutoff 25 January 2013)
Time Frame: Screening Visit, Every 8 weeks (or 9 weeks if receiving topotecan) until progression reported between day of first participant randomized (29 October 2009) until cutoff date of 25 January 2013
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 182 | 179
percentage of participants | 75.8 | 71.5

5. Primary Outcome: Progression Free Survival (PFS; Data Cutoff 14 November 2011)
Description: PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the investigators according to the RECIST criteria (for participants with measurable disease), and for those with non-measurable disease presence or absence of lesions was noted. Time from randomization to occurrence of disease progression or death was measured in months. An event was defined as the earliest progressive disease or death that occurred on or before the cutoff date (14 November 2011), regardless of start of nonprotocol specified anti-cancer therapy or the bevacizumab monotherapy. Disease progression was assessed by investigator according to RECIST or by symptom deterioration, and could not be declared on the basis of rising cancer antigen 125 (CA125) levels alone. Kaplan-Meier methodology was used. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: ITT Population; only participants with an event of progression or death were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 168 | 141
months | 3.4 [2.10 to 3.75] | 6.8 [5.62 to 7.79]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.379, 95% CI 2-sided [0.296 to 0.485] — Stratified analysis:Strata were chemotherapy selected (paclitaxel, PLD, or topotecan), prior anti-angiogenic therapy (yes or no), and platinum-free interval (less than [<] 3 or 3-6 months). Cox regression model was used to determine the hazard ratio
Statistical Analysis 2: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p < 0.0001, Log Rank; Unstratified analysis; Hazard Ratio (HR) = 0.460, 95% CI 2-sided [0.366 to 0.577]
Statistical Analysis 3: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p < 0.0001, Peto-Peto-Prentice; Unstratified analysis
Statistical Analysis 4: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p < 0.0001, Peto-Peto-Prentice; Stratified analysis:Strata were chemotherapy selected, prior anti-angiogenic therapy, and platinum-free interval

6. Secondary Outcome: Overall Survival (Data Cutoff 25 January 2013)
Description: Duration of overall survival was defined as the time from randomization to death of any cause. Kaplan-Meier methodology was used. The OS data for participants for whom no death was captured in the clinical database were censored at the last time they were known to be alive. 95% CI was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 4
Population: ITT Population; only participants who died were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 138 | 128
months | 13.3 [11.89 to 16.43] | 16.6 [13.70 to 18.99]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.1360, Log Rank — Unstratified analysis; Hazard Ratio (HR) = 0.833, 95% CI 2-sided [0.655 to 1.059]
Statistical Analysis 2: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.0715, Peto-Peto-Prentice — Unstratified analysis
Statistical Analysis 3: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.2711, Log Rank — [p-value comment as in outcome 2, analysis 3]; Hazard Ratio (HR) = 0.870, 95% CI 2-sided [0.678 to 1.116]
Statistical Analysis 4: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.0890, Peto-Peto-Prentice — [p-value comment as in outcome 2, analysis 3]

7. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Ovarian (OV) 28 Abdominal/Gastrointestinal (AB/GI) Symptom Scale - Percentage of Responders (Data Cutoff 14 November 2011)
Description: The EORTC OV-28 module is a questionnaire that focuses on issues specific to ovarian cancer. It assesses AB/GI symptoms, among others. Participants were asked to indicate the extent to which they experienced AB/GI symptoms in the week prior to assessment. Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) to the following: Did you have abdominal pain? Did you have a bloated feeling in your abdomen/stomach? Did you have problems with your clothes feeling too tight? Did you experience any change in bowel habit as a result of your disease or treatment? Were you troubled by passing wind/gas/flatulence? Have you felt full too quickly after beginning to eat? Have you had indigestion/heartburn? Data are transformed to a scale from 0 to 100. Lower scores represent better health (fewer symptoms). Participants were considered a responder if they had a 10 point or more reduction in EORTC QLQ-OV28 AB/GI symptom scale score from baseline.
Time Frame: Baseline and Weeks 8, 9, 16, 18, 24 and 30 (Data Cutoff 14 November 2011)
Population: ITT population; n (number) = (equals) number of participants that completed the questionnaire at baseline and at the specified visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 84 | 122
percentage of participants
  Weeks 8/9 | 19.0 [11.3 to 29.1] | 27.9 [20.1 to 36.7]
  Weeks 16/18: number analyzed (Participants) | 43 | 86
  Weeks 16/18 | 23.3 [11.8 to 38.6] | 26.7 [17.8 to 37.4]
  Week 24: number analyzed (Participants) | 22 | 53
  Week 24 | 22.7 [7.8 to 45.4] | 32.1 [19.9 to 46.3]
  Week 30: number analyzed (Participants) | 12 | 42
  Week 30 | 33.3 [9.9 to 65.1] | 28.6 [15.7 to 44.6]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Comparison of responders at baseline versus Week 8/9; Test type: Superiority or Other; p = 0.1859, Fisher Exact; Difference in Response Rates = 8.8, 95% CI 2-sided [-3.8 to 21.4] — 95% CI was approximated with Hauck-Anderson continuity correction
Statistical Analysis 2: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Comparison of responders at baseline versus at Week 16/18; Test type: Superiority or Other; p = 0.8309, Fisher Exact; Difference in Response Rates = 3.5, 95% CI 2-sided [-14 to 20.9] — 95% CI was approximated with Hauck-Anderson continuity correction
Statistical Analysis 3: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Comparison of responders at baseline versus at Week 24; Test type: Superiority or Other; p = 0.5790, Fisher Exact; Difference in Response Rates = 9.3, 95% CI 2-sided [-15 to 34.1] — 95% CI was approximated with Hauck-Anderson continuity correction
Statistical Analysis 4: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Comparison of responders at baseline versus at Week 30; Test type: Superiority or Other; p = 0.7339, Fisher Exact; Difference in Response Rates = -4.8, 95% CI 2-sided [-40 to 30.6] — 95% CI was approximated with Hauck-Anderson continuity correction

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were recorded at every treatment visit and all follow-up visits until 2 months after the final follow-up visit (up to approximately 4 years).
Description: Only Grade 2-5 AEs according to National Cancer Institute Common Terminology Criteria for AEs (NCI-CTCAE) were recorded per the protocol. The safety population included all treated participants.
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 49/181 | 56/179
Other Adverse Events (participants affected / at risk) | 129/181 | 146/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=181) | Chemotherapy + Bevacizumab (N=179)
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Ileus (Gastrointestinal disorders) | 2 | 4
Subileus (Gastrointestinal disorders) | 6 | 4
Constipation (Gastrointestinal disorders) | 2 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 7 | 0
General physical health deterioration (General disorders) | 1 | 3
Pyrexia (General disorders) | 3 | 3
Fatigue (General disorders) | 2 | 0
Device related infection (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Vesical fistula (Renal and urinary disorders) | 0 | 2
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Hypertension (Vascular disorders) | 0 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Haemorrhagic ascites (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Catheter site necrosis (General disorders) | 0 | 1
General symptom (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infectious peritonitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Wrong drug administered (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Cytoreductive surgery (Surgical and medical procedures) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=181) | Chemotherapy + Bevacizumab (N=179)
Anaemia (Blood and lymphatic system disorders) | 46 | 35
Leukopenia (Blood and lymphatic system disorders) | 25 | 23
Neutropenia (Blood and lymphatic system disorders) | 44 | 55
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 10
Abdominal pain (Gastrointestinal disorders) | 15 | 17
Abdominal pain upper (Gastrointestinal disorders) | 4 | 9
Constipation (Gastrointestinal disorders) | 17 | 13
Diarrhoea (Gastrointestinal disorders) | 10 | 17
Nausea (Gastrointestinal disorders) | 13 | 17
Vomiting (Gastrointestinal disorders) | 15 | 14
Fatigue (General disorders) | 46 | 49
Mucosal inflammation (General disorders) | 10 | 23
Infection (Infections and infestations) | 6 | 19
Urinary tract infection (Infections and infestations) | 13 | 15
Weight decreased (Investigations) | 5 | 11
Decreased appetite (Metabolism and nutrition disorders) | 14 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 13 | 32
Proteinuria (Renal and urinary disorders) | 1 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 15
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 | 19
Hypertension (Vascular disorders) | 10 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.